CLINICAL TRIAL: NCT02214160
Title: An Open-label Long-Term Safety and Efficacy Extension Study in Subjects With Long-Chain Fatty Acid Oxidation Disorders (LC-FAOD) Previously Enrolled in UX007 or Triheptanoin Studies
Brief Title: Long-Chain Fatty Acid Oxidation Disorders (LC-FAOD) Extension Study for Subjects Previously Enrolled in Triheptanoin Studies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UX007-CL202; 2016-000322-19 (EudraCT Number)
Expanded Access: NCT03773770 (Available)
Record Dates: First submitted 2014-08-06; First posted 2014-08-12 (Estimated); Results first posted 2021-12-08 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Carnitine Palmitoyltransferase (CPT I or CPT II) Deficiency; Very Long Chain Acyl-CoA Dehydrogenase (VLCAD) Deficiency; Long-chain 3-hydroxy-acyl-CoA Dehydrogenase (LCHAD) Deficiency; Trifunctional Protein (TFP) Deficiency; Carnitine-acylcarnitine Translocase (CACT) Deficiency
Keywords: Long-Chain Fatty Acid Oxidation Disorders (LC-FAOD); carnitine palmitoyltransferase (CPT I or CPT II) deficiency; very long chain acyl-CoA dehydrogenase (VLCAD) deficiency; long-chain 3-hydroxy-acyl-CoA dehydrogenase (LCHAD) deficiency; trifunctional protein (TFP) deficiency; carnitine-acylcarnitine translocase (CACT) deficiency; Triheptanoin; UX007; C7
MeSH Terms: conditions — VLCAD deficiency | interventions — triheptanoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- UX007 (Experimental): Participants previously treated with UX007 or treatment-naive participants will begin or continue treatment with daily open-label UX007 while maintaining their other dietary restrictions.
  Interventions: Drug: UX007

INTERVENTIONS:
Drug: UX007 — Administered orally (PO) with food or by gastrostomy tube, at the target dose range of 25-35% of total calories.
  Other Names: Triheptanoin; C7

SUMMARY:
The primary objective of this study is to evaluate the long-term safety and efficacy of UX007 in participants with LC-FAOD. The secondary objectives of this study are to evaluate the effect of UX007 on energy metabolism in LC-FAOD and evaluate the impact of UX007 on clinical events associated with LC-FAOD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 6 months of age or older
2. Prior participation in a clinical study assessing UX007/triheptanoin treatment for LC FAOD. Study Sponsors/Collaborators include: Oregon Health & Science University, University of Pittsburgh, and Ultragenyx Pharmaceutical (ClinicalTrials.gov Identifiers: NCT01379625, NCT01461304, and NCT01886378). Patients who received UX007/triheptanoin treatment as part of other clinical studies; investigator sponsored trials (IST); expanded access/compassionate use treatment programs; or patients who are treatment naïve (i.e., naïve to both UX007 and food-grade triheptanoin), have failed conventional therapy and, in the opinion of the Investigator and Sponsor, have documented clear unmet need, may also be eligible at the discretion of the Sponsor
3. Confirmed diagnosis of LC-FAOD including: CPT I or CPT II deficiency, VLCAD deficiency, LCHAD deficiency, TFP deficiency, or CACT deficiency. Information on diagnosis will be obtained from medical records and should include confirmed diagnosis by results of acylcarnitine profiles, fatty acid oxidation probe studies in cultured fibroblasts, and/or mutation analysis
4. Willing and able to complete all aspects of the study through the end of the study, including visits and tests, documentation of symptoms and diet, and administration of study medications. If a minor, have a caregiver(s) willing and able to assist in all applicable study requirements
5. Provide written informed consent (subjects aged ≥ 18 years), or provide written assent (where appropriate) and have a legally authorized representative willing and able to provide written informed consent, after the nature of the study has been explained and prior to any research-related procedures.
6. Females of child-bearing potential must have a negative urine pregnancy test at Baseline and be willing to have additional pregnancy tests during the study. Females considered not of child-bearing potential include those who have not experienced menarche, are post-menopausal (defined as having no menses for at least 12 months without an alternative medical cause), or are permanently sterile due to total hysterectomy, bilateral salpingectomy, or bilateral oophorectomy
7. Participants of child-bearing potential or fertile males with partners of child-bearing potential who are sexually active must consent to use a highly effective method of contraception as determined by the Investigator from the period following the signing of the informed consent through 30 days after last dose of study drug

Exclusion Criteria:

1. Diagnosis of medium-chain acyl coenzyme A dehydrogenase (MCAD) deficiency, short- or medium-chain FAOD, ketone body metabolism defect, propionic acidemia or methylmalonic acidemia
2. Patient qualifies for any other clinical trial designed to progressively evaluate the safety and efficacy of triheptanoin in LC-FAOD
3. Any known hypersensitivity to triheptanoin that, in the judgment of the Investigator, places the subject at increased risk for adverse effects
4. Pregnant and/or breastfeeding an infant at Screening or planning to become pregnant (self or partner) at any time during the study
5. Have any co-morbid conditions, including unstable major organ-system disease(s) that in the opinion of the Investigator, places the subject at increased risk of complications, interferes with study participation or compliance, or confounds study objectives, or unwilling to discontinue prohibited medications

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2014-12-09 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Inc.
Locations (11):
- United States (9):
  - University of California San Francisco, San Francisco, California
  - Children's National Health System, Washington D.C., District of Columbia
  - University of South Florida, Tampa, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Vanderbilt Medical Center, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- United Kingdom (2):
  - National Hospital for Neurology and Neurosurgery, London
  - Great Ormond Street Hospital, London

REFERENCES:
- [Background] Vockley J, Burton B, Berry G, Longo N, Phillips J, Sanchez-Valle A, Chapman K, Tanpaiboon P, Grunewald S, Murphy E, Lu X, Cataldo J. Effects of triheptanoin (UX007) in patients with long-chain fatty acid oxidation disorders: Results from an open-label, long-term extension study. J Inherit Metab Dis. 2021 Jan;44(1):253-263. doi: 10.1002/jimd.12313. Epub 2020 Sep 14. PMID 32885845
- [Background] Vockley J, Burton BK, Berry G, Longo N, Phillips J, Sanchez-Valle A, Chapman KA, Tanpaiboon P, Grunewald S, Murphy E, Lu X, Rahman S, Ray K, Reineking B, Pisani L, Ramirez AN. Triheptanoin for the treatment of long-chain fatty acid oxidation disorders: Final results of an open-label, long-term extension study. J Inherit Metab Dis. 2023 Sep;46(5):943-955. doi: 10.1002/jimd.12640. Epub 2023 Jun 19. PMID 37276053

RESULTS

PARTICIPANT FLOW:
Groups:
- UX007-CL201-Rollover Cohort: Participants who participated in the UX007-CL201 study (NCT01886378) receive UX007, administered orally with food or by gastronomy tube (usually 4 times per day: breakfast, lunch, dinner, and before bed), at the target dose range of 25-35% of total calories.
- IST/Other Cohort: Participants who were previously treated with UX007/triheptanoin (including food-grade triheptanoin) in an investigator sponsored trial (IST) or another UX007/triheptanoin study receive UX007, administered orally with food or by gastronomy tube (usually 4 times per day: breakfast, lunch, dinner, and before bed), at the target dose range of 25-35% of total calories.
- Triheptanoin-Naïve Cohort: Participants who are UX007 treatment-naïve (i.e., naïve to both UX007 and food-grade triheptanoin), or who had failed conventional therapy (including those who participated in UX007-CL201 study previously but were off UX007 for more than 2 years preceding enrollment into CL202) receive UX007, administered orally with food or by gastronomy tube (usually 4 times per day: breakfast, lunch, dinner, and before bed), at the target dose range of 25-35% of total calories.
Period: Overall Study
Arm/Group | UX007-CL201-Rollover Cohort | IST/Other Cohort | Triheptanoin-Naïve Cohort
Started | 24 | 37 | 33
Completed | 20 | 29 | 23
Not Completed | 4 | 8 | 10
Not completed — Withdrawal by Subject | 1 | 0 | 6
Not completed — Death | 2 | 2 | 1
Not completed — Subject Non-Compliance | 0 | 3 | 1
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Sponsor Decision | 0 | 2 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | UX007-CL201-Rollover Cohort | IST/Other Cohort | Triheptanoin-Naïve Cohort | Total
Number analyzed (Participants) | 24 | 37 | 33 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.16 (14.310) | 17.69 (14.490) | 9.33 (9.745) | 13.60 (13.333)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 21 | 14 | 45
  Male | 14 | 16 | 19 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 5 | 12
  Not Hispanic or Latino | 21 | 30 | 28 | 79
  Unknown or Not Reported | 0 | 3 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 1 | 3
  Black or African American | 1 | 1 | 2 | 4
  White | 21 | 33 | 28 | 82
  Other, Not Specified | 1 | 2 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Annualized LC-FAOD Major Clinical Events (MCEs) Rate: 18 Months Pre- and Entire UX007 Period Comparison for UX007-CL201-Rollover Cohort
Description: The annualized LC-FAOD MCE rate, inclusive of skeletal myopathy (rhabdomyolysis), hepatic (hypoglycemia) and cardiomyopathy events, defined as any visit to the emergency room (ER)/acute care, hospitalization, emergency intervention (i.e. any unscheduled administration of therapeutics at home or in the clinic), or any similar event whether caused primarily by LC-FAOD or by an intercurrent illness complicated by LC-FAOD.
  The annualized event rate was calculated at the number of events divided by the duration of data collection period in days/365.25
Time Frame: Pre-UX007 treatment period (up to 18 months) and post-UX007 treatment period (up to 2072 days)
Population: Full Analysis Set: all participants enrolled who had at least 1 post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: events/year
Arm/Group | UX007-CL201-Rollover Cohort
Number analyzed (Participants) | 24
events/year
  Pre-UX007 Period | 1.76 (1.64)
  UX007 Treatment Period | 1.00 (1.00)
Statistical Analysis 1: Comparison: UX007-CL201-Rollover Cohort; Test type: Superiority; p = 0.0347, Paired T-test

2. Primary Outcome: Annualized LC-FAOD MCEs Rate: 18 Months Pre- and Entire UX007 Period Comparison for IST/Other Cohort and Triheptanoin-Naïve Cohort
Description: as for outcome 1
Time Frame: Pre-UX007 treatment period (up to 18 months) and post-UX007 treatment period (up to 2072 days)
Population: Full Analysis Set: all participants enrolled who had at least 1 post-baseline efficacy assessment. Per protocol, pre-UX007 MCE data was not collected in the IST/Other Cohort.
Measure: Median (Inter-Quartile Range); unit: events/year
Arm/Group | IST/Other Cohort | Triheptanoin-Naïve Cohort
Number analyzed (Participants) | 37 | 33
events/year
  Pre-UX007 Period: number analyzed (Participants) | 0 | 33
  Pre-UX007 Period |  | 2.00 [0.67 to 3.33]
  UX007 Treatment Period | 0.57 [0.0 to 1.67] | 0.28 [0.00 to 1.43]
Statistical Analysis 1: Comparison: Triheptanoin-Naïve Cohort; Test type: Superiority; p = 0.0343, Wilcoxon Signed Rank Test

3. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) or Serious TEAEs
Description: An adverse event (AE) was defined as any untoward medical occurrence, whether or not considered drug related. A serious adverse event (SAE) results in any of the following outcomes: death; a life-threatening AE; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant incapacity or disability; a congenital anomaly/birth defect; an important medical event. AEs were graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 (mild=1, moderate=2, severe=3, life-threatening=4, death=5).
Time Frame: Post-UX007 treatment through the end of treatment (up to 2072 days) plus 30-35 days
Population: Safety Analysis Set: participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | UX007-CL201-Rollover Cohort | IST/Other Cohort | Triheptanoin-Naïve Cohort
Number analyzed (Participants) | 24 | 37 | 33
participants
  >= 1 TEAE | 24 | 35 | 32
  Treatment-Related TEAEs | 14 | 22 | 28
  Treatment-Related Gastrointestinal (GI) TEAEs | 10 | 19 | 27
  Grade 3 TEAEs | 16 | 26 | 18
  Grade 4 TEAEs | 3 | 2 | 2
  Serious TEAEs | 20 | 28 | 22
  Treatment-Related Serious TEAEs | 1 | 1 | 3
  TEAEs Leading to Treatment Discontinuation | 1 | 1 | 1
  TEAEs Leading to Study Discontinuation | 0 | 1 | 1
  TEAEs Leading to Death | 2 | 2 | 1

4. Secondary Outcome: Change From Baseline in Echocardiogram (ECHO) Parameters Over Time: Left Ventricular Mass Index (LVMI)
Time Frame: Baseline, Month 12, Month 24, Month 36, Month 48, Month 60
Population: Full Analysis Set: all participants enrolled who had at least 1 post-baseline efficacy assessment. Participants with a value at baseline and given time point.
Measure: Mean (Standard Deviation); unit: g/m
Arm/Group | UX007-CL201-Rollover Cohort | IST/Other Cohort | Triheptanoin-Naïve Cohort
Number analyzed (Participants) | 24 | 37 | 33
g/m
  Change at Month 12: number analyzed (Participants) | 15 | 29 | 16
  Change at Month 12 | -5.27 (21.433) | 4.55 (21.903) | -9.06 (29.965)
  Change at Month 24: number analyzed (Participants) | 11 | 27 | 9
  Change at Month 24 | -2.73 (23.711) | -0.37 (18.132) | 1.00 (39.459)
  Change at Month 36: number analyzed (Participants) | 12 | 26 | 6
  Change at Month 36 | -6.75 (28.933) | 1.23 (19.488) | 12.33 (38.831)
  Change at Month 48: number analyzed (Participants) | 3 | 23 | 3
  Change at Month 48 | -12.33 (29.263) | -1.04 (21.900) | -9.67 (36.529)
  Change at Month 60: number analyzed (Participants) | 0 | 6 | 0
  Change at Month 60 |  | 8.83 (25.639) |

5. Secondary Outcome: Change From Baseline in ECHO Parameters Over Time: Left Ventricular Mass (LVM)
Time Frame: Baseline, Month 12, Month 24, Month 36, Month 48, Month 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: g
Groups:
- Triheptanoin-Naïve Cohort: Participants who are UX007 treatment-naïve (i.e., naïve to both UX007 and food-grade triheptanoin), or who had failed conventional therapy (including those who participated in UX007-CL201 study previously but were off UX007 for more than 2 years preceding enrollment into CL202) receive UX007, administered orally with food or by gastronomy tube (usually 4 times per day: breakfast, lunch, dinner, and before bed), at the target dose range of 25-35% of total calories.
  -
Arm/Group | UX007-CL201-Rollover Cohort | IST/Other Cohort | Triheptanoin-Naïve Cohort
Number analyzed (Participants) | 24 | 37 | 33
g
  Change at Month 12: number analyzed (Participants) | 18 | 31 | 20
  Change at Month 12 | -1.50 (29.374) | 12.58 (22.648) | -0.75 (25.935)
  Change at Month 24: number analyzed (Participants) | 17 | 28 | 12
  Change at Month 24 | 9.71 (27.034) | 5.61 (34.465) | 3.25 (38.833)
  Change at Month 36: number analyzed (Participants) | 14 | 28 | 8
  Change at Month 36 | 6.21 (30.355) | 16.36 (36.898) | 15.75 (48.922)
  Change at Month 48: number analyzed (Participants) | 4 | 25 | 4
  Change at Month 48 | 33.25 (12.842) | 19.72 (42.645) | 10.25 (52.753)
  Change at Month 60: number analyzed (Participants) | 0 | 7 | 0
  Change at Month 60 |  | 46.29 (19.102) |

6. Secondary Outcome: Change From Baseline in ECHO Parameters Over Time: Left Ventricular Diameter (LVD)
Time Frame: Baseline, Month 12, Month 24, Month 36, Month 48, Month 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | UX007-CL201-Rollover Cohort | IST/Other Cohort | Triheptanoin-Naïve Cohort
Number analyzed (Participants) | 24 | 37 | 33
mm
  Change at Month 12: number analyzed (Participants) | 18 | 29 | 21
  Change at Month 12 | 2.19 (9.138) | 2.38 (8.719) | 1.57 (4.308)
  Change at Month 24: number analyzed (Participants) | 17 | 27 | 12
  Change at Month 24 | 3.26 (11.158) | 3.00 (8.535) | 0.67 (4.755)
  Change at Month 36: number analyzed (Participants) | 17 | 26 | 9
  Change at Month 36 | -0.11 (13.174) | 3.23 (8.883) | 4.78 (5.094)
  Change at Month 48: number analyzed (Participants) | 4 | 23 | 5
  Change at Month 48 | 10.88 (17.264) | 3.82 (9.115) | 2.60 (5.177)
  Change at Month 60: number analyzed (Participants) | 0 | 7 | 1
  Change at Month 60 |  | 40.29 (5.407) | 50.00 (NA) — 1 participant at this time point

7. Secondary Outcome: Change From Baseline in ECHO Parameters Over Time: Left Ventricular Ejection Fraction (LVEF)
Time Frame: Baseline, Month 12, Month 18, Month 24, Month 30, Month 36, Month 48, Month 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent of blood ejected during systole
Arm/Group | UX007-CL201-Rollover Cohort | IST/Other Cohort | Triheptanoin-Naïve Cohort
Number analyzed (Participants) | 24 | 37 | 33
percent of blood ejected during systole
  Change at Month 12: number analyzed (Participants) | 21 | 31 | 21
  Change at Month 12 | 0.76 (7.602) | 1.32 (7.254) | 0.71 (6.474)
  Change at Month 18: number analyzed (Participants) | 0 | 0 | 1
  Change at Month 18 |  |  | 0.00 (NA) — 1 participant at this time point
  Change at Month 24: number analyzed (Participants) | 22 | 25 | 13
  Change at Month 24 | -1.86 (9.062) | 0.24 (8.875) | 2.31 (8.400)
  Change at Month 30: number analyzed (Participants) | 1 | 0 | 0
  Change at Month 30 | 0.00 (NA) — 1 participant at this time point |  |
  Change at Month 36: number analyzed (Participants) | 21 | 26 | 9
  Change at Month 36 | -1.10 (7.259) | -1.92 (5.986) | 3.44 (7.601)
  Change at Month 48: number analyzed (Participants) | 6 | 23 | 5
  Change at Month 48 | -1.33 (3.445) | -1.57 (7.464) | 1.60 (5.459)
  Change at Month 60: number analyzed (Participants) | 0 | 7 | 1
  Change at Month 60 |  | -5.00 (7.394) | 1.00 (NA) — 1 participant at this time point

8. Secondary Outcome: Change From Baseline in ECHO Parameters Over Time: LVEF Z-Score (Pediatric Participants)
Description: The Z-scores express the deviation (or how far away) the measure is from the mean LVEF based on the size or age of the pediatric participants:
  Z-score=0 indicates the participant is exactly the same as the mean of the healthy general population.
  Z-score=-1 indicates it's 1 standard deviation below the mean of the healthy population.
  Z-score=+1 indicates it's 1 standard deviation above the mean.
Time Frame: Baseline, Month 12, Month 24, Month 36
Population: Full Analysis Set: all participants enrolled who had at least 1 post-baseline efficacy assessment. Pediatric participants with a value at baseline and given time point.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | UX007-CL201-Rollover Cohort | IST/Other Cohort | Triheptanoin-Naïve Cohort
Number analyzed (Participants) | 5 | 1 | 8
Z-score
  Change at Month 12: number analyzed (Participants) | 4 | 1 | 4
  Change at Month 12 | 0.34 (1.229) | 1.84 (NA) — 1 participant at this time point | 0.21 (1.492)
  Change at Month 24: number analyzed (Participants) | 4 | 1 | 2
  Change at Month 24 | -0.05 (1.469) | 2.28 (NA) — 1 participant at this time point | 0.72 (1.103)
  Change at Month 36: number analyzed (Participants) | 0 | 1 | 1
  Change at Month 36 |  | -0.52 (NA) — 1 participant at this time point | -0.66 (NA) — 1 participant at this time point

9. Secondary Outcome: Change From Baseline in ECHO Parameters Over Time: Left Ventricular Shortening Fraction (LVSF)
Description: Fractional shortening is calculated by measuring the percentage change in left ventricular diameter during systole. A negative value indicates less ventricular/muscular contractility, and a positive value indicates more ventricular/muscular contractility.
Time Frame: Baseline, Month 12, Month 24, Month 30, Month 36, Month 48, Month 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: % change in left ventricular diameter
Arm/Group | UX007-CL201-Rollover Cohort | IST/Other Cohort | Triheptanoin-Naïve Cohort
Number analyzed (Participants) | 24 | 37 | 33
% change in left ventricular diameter
  Change at Month 12: number analyzed (Participants) | 20 | 32 | 21
  Change at Month 12 | -1.30 (5.564) | -0.91 (6.468) | -1.48 (5.904)
  Change at Month 24: number analyzed (Participants) | 20 | 29 | 14
  Change at Month 24 | -1.90 (6.052) | 1.03 (6.242) | -1.36 (7.967)
  Change at Month 30: number analyzed (Participants) | 1 | 0 | 0
  Change at Month 30 | -7.00 (NA) — 1 participant at this time point |  |
  Change at Month 36: number analyzed (Participants) | 20 | 28 | 9
  Change at Month 36 | -0.10 (6.086) | 0.25 (4.502) | 1.11 (5.395)
  Change at Month 48: number analyzed (Participants) | 4 | 25 | 5
  Change at Month 48 | 3.00 (4.320) | 0.52 (4.501) | -0.60 (6.269)
  Change at Month 60: number analyzed (Participants) | 0 | 7 | 1
  Change at Month 60 |  | -0.57 (4.392) | 0.00 (NA) — 1 participant at this time point

10. Secondary Outcome: Change From Baseline in ECHO Parameters Over Time: LVSF Z-Score (Pediatric Participants)
Description: The Z-scores express the deviation (or how far away) the measure is from the mean LVSF based on the size or age of the pediatric participants:
  Z-score=0 indicates the participant is exactly the same as the mean of the healthy general population.
  Z-score=-1 indicates it's 1 standard deviation below the mean of the healthy population.
  Z-score=+1 indicates it's 1 standard deviation above the mean.
Time Frame: Baseline, Month 12, Month 24, Month 36, Month 48, Month 60
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | UX007-CL201-Rollover Cohort | IST/Other Cohort | Triheptanoin-Naïve Cohort
Number analyzed (Participants) | 24 | 37 | 33
Z-score
  Change at Month 12: number analyzed (Participants) | 11 | 25 | 14
  Change at Month 12 | 0.10 (1.659) | 0.25 (1.315) | -0.38 (1.597)
  Change at Month 24: number analyzed (Participants) | 11 | 23 | 9
  Change at Month 24 | 0.27 (2.255) | 0.30 (1.607) | 0.13 (2.119)
  Change at Month 36: number analyzed (Participants) | 7 | 23 | 8
  Change at Month 36 | 0.75 (1.729) | 0.13 (1.115) | 0.58 (1.943)
  Change at Month 48: number analyzed (Participants) | 3 | 20 | 5
  Change at Month 48 | 0.53 (0.316) | 0.24 (1.464) | 0.10 (1.888)
  Change at Month 60: number analyzed (Participants) | 0 | 6 | 0
  Change at Month 60 |  | -0.45 (0.834) |

11. Secondary Outcome: Annualized Duration Rate of All MCEs
Description: The annualized duration rate of LC-FAOD MCEs, inclusive of skeletal myopathy (rhabdomyolysis), hepatic (hypoglycemia) and cardiomyopathy events, and defined as any visit to the ER/acute care, hospitalization, emergency intervention (i.e. any unscheduled administration of therapeutics at home or in the clinic), or any similar event whether caused primarily by LC-FAOD or by an intercurrent illness complicated by LC-FAOD. The annualized duration rate is calculated as the total duration (days) of events divided by the duration of data collection period in days/365.25.
Time Frame: Post-UX007 treatment through the end of the study (up to 2072 days)
Population: Full Analysis Set: all participants enrolled who had at least 1 post-baseline efficacy assessment.
Measure: Median (Inter-Quartile Range); unit: days/year
Arm/Group | UX007-CL201-Rollover Cohort | IST/Other Cohort | Triheptanoin-Naïve Cohort
Number analyzed (Participants) | 24 | 37 | 33
days/year | 2.123 [0.000 to 9.766] | 2.487 [0.000 to 6.968] | 0.796 [0.000 to 5.484]

12. Secondary Outcome: Annualized Event Rate of Rhabdomyolysis MCEs
Description: The annualized event rate of LC-FAOD major events of skeletal myopathy (rhabdomyolysis), defined as any visit to the ER/acute care, hospitalization, emergency intervention (i.e. any unscheduled administration of therapeutics at home or in the clinic), or any similar event whether caused primarily by LC-FAOD or by an intercurrent illness complicated by LC-FAOD.
  The annualized event rate was calculated at the number of events divided by the duration of data collection period in days/365.25.
Time Frame: Post-UX007 treatment through the end of the study (up to 2072 days)
Population: Full Analysis Set: all participants enrolled who had at least 1 post-baseline efficacy assessment.
Measure: Median (Inter-Quartile Range); unit: events/year
Arm/Group | UX007-CL201-Rollover Cohort | IST/Other Cohort | Triheptanoin-Naïve Cohort
Number analyzed (Participants) | 24 | 37 | 33
events/year | 0.352 [0.000 to 1.472] | 0.574 [0.000 to 1.673] | 0.281 [0.000 to 1.425]

13. Secondary Outcome: Annualized Duration Rate of Rhabdomyolysis MCEs
Description: The annualized duration rate of LC-FAOD skeletal myopathy (rhabdomyolysis) MCEs, defined as any visit to the ER/acute care, hospitalization, emergency intervention (i.e. any unscheduled administration of therapeutics at home or in the clinic), or any similar event whether caused primarily by LC-FAOD or by an intercurrent illness complicated by LC-FAOD.
  The annualized duration rate is calculated as the total duration (days) of events divided by the duration of data collection period in days/365.25.
Time Frame: Post-UX007 treatment through the end of the study (up to 2072 days)
Population: Full Analysis Set: all participants enrolled who had at least 1 post-baseline efficacy assessment.
Measure: Median (Inter-Quartile Range); unit: days/year
Arm/Group | UX007-CL201-Rollover Cohort | IST/Other Cohort | Triheptanoin-Naïve Cohort
Number analyzed (Participants) | 24 | 37 | 33
days/year | 2.123 [0.000 to 6.969] | 2.487 [0.000 to 6.948] | 0.448 [0.000 to 5.398]

14. Secondary Outcome: Annualized Event Rate of Cardiomyopathy MCEs
Description: The annualized event rate of LC-FAOD major events inclusive of cardiomyopathy events, defined as any visit to the ER/acute care, hospitalization, emergency intervention (i.e. any unscheduled administration of therapeutics at home or in the clinic), or any similar event whether caused primarily by LC-FAOD or by an intercurrent illness complicated by LC-FAOD.
  The annualized event rate was calculated at the number of events divided by the duration of data collection period in days/365.25.
Time Frame: Post-UX007 treatment through the end of the study (up to 2072 days)
Population: Full Analysis Set: all participants enrolled who had at least 1 post-baseline efficacy assessment.
Measure: Median (Inter-Quartile Range); unit: event/year
Arm/Group | UX007-CL201-Rollover Cohort | IST/Other Cohort | Triheptanoin-Naïve Cohort
Number analyzed (Participants) | 24 | 37 | 33
event/year | 0.000 [0.000 to 0.120] | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]

15. Secondary Outcome: Annualized Duration Rate of Cardiomyopathy MCEs
Description: The annualized duration rate of LC-FAOD cardiomyopathy MCEs, defined as any visit to the ER/acute care, hospitalization, emergency intervention (i.e. any unscheduled administration of therapeutics at home or in the clinic), or any similar event whether caused primarily by LC-FAOD or by an intercurrent illness complicated by LC-FAOD.
  The annualized duration rate is calculated as the total duration (days) of events divided by the duration of data collection period in days/365.25
Time Frame: Post-UX007 treatment through the end of the study (up to 2072 days)
Population: Full Analysis Set: all participants enrolled who had at least 1 post-baseline efficacy assessment.
Measure: Median (Inter-Quartile Range); unit: days/year
Arm/Group | UX007-CL201-Rollover Cohort | IST/Other Cohort | Triheptanoin-Naïve Cohort
Number analyzed (Participants) | 24 | 37 | 33
days/year | 0.000 [0.000 to 0.174] | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]

16. Secondary Outcome: Annualized Event Rate of Hypoglycemic MCEs
Description: The annualized event rate of LC-FAOD major events of hepatic (hypoglycemia) events, defined as any visit to the ER/acute care, hospitalization, emergency intervention (i.e. any unscheduled administration of therapeutics at home or in the clinic), or any similar event whether caused primarily by LC-FAOD or by an intercurrent illness complicated by LC-FAOD.
  The annualized event rate was calculated at the number of events divided by the duration of data collection period in days/365.25.
Time Frame: Post-UX007 treatment through the end of the study (up to 2072 days)
Population: Full Analysis Set: all participants enrolled who had at least 1 post-baseline efficacy assessment.
Measure: Median (Inter-Quartile Range); unit: events/year
Arm/Group | UX007-CL201-Rollover Cohort | IST/Other Cohort | Triheptanoin-Naïve Cohort
Number analyzed (Participants) | 24 | 37 | 33
events/year | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]

17. Secondary Outcome: Annualized Duration Rate of Hypoglycemic MCEs
Description: The annualized duration rate of LC-FAOD hepatic (hypoglycemia) MCEs, defined as any visit to the ER/acute care, hospitalization, emergency intervention (i.e. any unscheduled administration of therapeutics at home or in the clinic), or any similar event whether caused primarily by LC-FAOD or by an intercurrent illness complicated by LC-FAOD.
  The annualized duration rate is calculated as the total duration (days) of events divided by the duration of data collection period in days/365.25.
Time Frame: Post-UX007 treatment through the end of the study (up to 2072 days)
Population: Full Analysis Set: all participants enrolled who had at least 1 post-baseline efficacy assessment.
Measure: Median (Inter-Quartile Range); unit: days/year
Arm/Group | UX007-CL201-Rollover Cohort | IST/Other Cohort | Triheptanoin-Naïve Cohort
Number analyzed (Participants) | 24 | 37 | 33
days/year | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]

ADVERSE EVENTS:
Time Frame: Post-UX007 treatment through the end of treatment (up to 2072 days) plus 30-35 days
Groups:
- All Participants: All participants received UX007, administered orally with food or by gastronomy tube (usually 4 times per day: breakfast, lunch, dinner, and before bed), at the target dose range of 25-35% of total calories.
Arm/Group | UX007-CL201-Rollover Cohort | IST/Other Cohort | Triheptanoin-Naïve Cohort | All Participants
All-Cause Mortality (participants affected / at risk) | 2/24 | 2/37 | 1/33 | 5/94
Serious Adverse Events (participants affected / at risk) | 20/24 | 28/37 | 22/33 | 70/94
Other Adverse Events (participants affected / at risk) | 24/24 | 34/37 | 32/33 | 90/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UX007-CL201-Rollover Cohort (N=24) | IST/Other Cohort (N=37) | Triheptanoin-Naïve Cohort (N=33) | All Participants (N=94)
ARRHYTHMIA (Cardiac disorders) | 1 | 0 | 0 | 1
CARDIAC ARREST (Cardiac disorders) | 0 | 1 | 0 | 1
CARDIAC FAILURE (Cardiac disorders) | 2 | 1 | 0 | 3
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 | 0 | 1 | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 | 0 | 1 | 2
CARDIOMYOPATHY (Cardiac disorders) | 4 | 1 | 0 | 5
CARDIOPULMONARY FAILURE (Cardiac disorders) | 0 | 0 | 1 | 1
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 2 | 0 | 0 | 2
LEFT VENTRICULAR HYPERTROPHY (Cardiac disorders) | 0 | 1 | 0 | 1
LONG QT SYNDROME (Cardiac disorders) | 0 | 1 | 0 | 1
MYOCARDITIS (Cardiac disorders) | 1 | 0 | 0 | 1
CHRONIC GASTRITIS (Gastrointestinal disorders) | 0 | 0 | 1 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 2 | 2 | 4
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0 | 1
GASTRITIS (Gastrointestinal disorders) | 0 | 1 | 0 | 1
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 3 | 6 | 2 | 11
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 0 | 1 | 1
ILEUS (Gastrointestinal disorders) | 1 | 0 | 0 | 1
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 | 0 | 1 | 1
RECTAL POLYP (Gastrointestinal disorders) | 0 | 1 | 0 | 1
STEATORRHOEA (Gastrointestinal disorders) | 0 | 1 | 0 | 1
VOLVULUS (Gastrointestinal disorders) | 1 | 0 | 0 | 1
VOMITING (Gastrointestinal disorders) | 2 | 4 | 5 | 11
PYREXIA (General disorders) | 0 | 0 | 1 | 1
CELLULITIS (Infections and infestations) | 0 | 0 | 1 | 1
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 | 1 | 0 | 1
CROUP INFECTIOUS (Infections and infestations) | 1 | 1 | 1 | 3
DEVICE RELATED INFECTION (Infections and infestations) | 0 | 1 | 0 | 1
DIVERTICULITIS (Infections and infestations) | 0 | 1 | 0 | 1
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0 | 1
GASTRITIS VIRAL (Infections and infestations) | 0 | 1 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 5 | 5 | 2 | 12
GASTROENTERITIS VIRAL (Infections and infestations) | 4 | 3 | 2 | 9
GASTROINTESTINAL VIRAL INFECTION (Infections and infestations) | 0 | 0 | 1 | 1
HERPES SIMPLEX (Infections and infestations) | 0 | 0 | 1 | 1
INFLUENZA (Infections and infestations) | 2 | 8 | 1 | 11
KLEBSIELLA BACTERAEMIA (Infections and infestations) | 0 | 0 | 1 | 1
KLEBSIELLA INFECTION (Infections and infestations) | 0 | 1 | 0 | 1
ORAL CANDIDIASIS (Infections and infestations) | 0 | 1 | 0 | 1
PARAINFLUENZAE VIRUS INFECTION (Infections and infestations) | 0 | 0 | 1 | 1
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 | 0 | 2 | 2
PNEUMONIA (Infections and infestations) | 1 | 1 | 0 | 2
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 1 | 0 | 0 | 1
PYELONEPHRITIS (Infections and infestations) | 0 | 2 | 0 | 2
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0 | 1
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 2 | 0 | 1 | 3
RHINOVIRUS INFECTION (Infections and infestations) | 0 | 2 | 0 | 2
SEPSIS (Infections and infestations) | 0 | 1 | 0 | 1
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 | 1 | 0 | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 0 | 1 | 1
TONSILLITIS (Infections and infestations) | 1 | 0 | 0 | 1
TRACHEITIS (Infections and infestations) | 1 | 0 | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 2 | 1 | 5
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0 | 1
VIRAL CARDIOMYOPATHY (Infections and infestations) | 1 | 0 | 0 | 1
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 2 | 1 | 5
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
AMMONIA INCREASED (Investigations) | 0 | 1 | 0 | 1
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 | 0 | 1 | 1
BRAIN NATRIURETIC PEPTIDE INCREASED (Investigations) | 0 | 1 | 0 | 1
INFLUENZA A VIRUS TEST POSITIVE (Investigations) | 0 | 2 | 0 | 2
TRANSAMINASES INCREASED (Investigations) | 0 | 0 | 1 | 1
ACIDOSIS (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 3 | 2 | 0 | 5
HYPERAMMONAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
HYPOPHAGIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
METABOLIC DISORDER (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
JOINT INSTABILITY (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 14 | 25 | 15 | 54
SCOLIOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
PLEOMORPHIC ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 | 1 | 0 | 1
HEADACHE (Nervous system disorders) | 1 | 0 | 0 | 1
ISCHAEMIC STROKE (Nervous system disorders) | 0 | 0 | 1 | 1
LETHARGY (Nervous system disorders) | 0 | 1 | 0 | 1
MIGRAINE (Nervous system disorders) | 0 | 1 | 0 | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 | 0 | 1 | 1
POLYNEUROPATHY (Nervous system disorders) | 1 | 0 | 0 | 1
SEIZURE (Nervous system disorders) | 1 | 0 | 0 | 1
ANXIETY (Psychiatric disorders) | 0 | 1 | 0 | 1
LISTLESS (Psychiatric disorders) | 0 | 1 | 0 | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 | 1 | 0 | 3
RENAL FAILURE (Renal and urinary disorders) | 1 | 0 | 0 | 1
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
CHRONIC RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 3
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 4
TONSILLAR HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
ELECTIVE PROCEDURE (Surgical and medical procedures) | 1 | 0 | 0 | 1
HEART TRANSPLANT (Surgical and medical procedures) | 1 | 0 | 0 | 1
HAEMODYNAMIC INSTABILITY (Vascular disorders) | 1 | 0 | 0 | 1
POOR VENOUS ACCESS (Vascular disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | UX007-CL201-Rollover Cohort (N=24) | IST/Other Cohort (N=37) | Triheptanoin-Naïve Cohort (N=33) | All Participants (N=94)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1 | 2 | 3
CARDIOMYOPATHY (Cardiac disorders) | 3 | 3 | 1 | 7
PALPITATIONS (Cardiac disorders) | 2 | 0 | 0 | 2
EAR PAIN (Ear and labyrinth disorders) | 2 | 0 | 1 | 3
MOTION SICKNESS (Ear and labyrinth disorders) | 0 | 0 | 3 | 3
ASTIGMATISM (Eye disorders) | 1 | 0 | 2 | 3
HYPERMETROPIA (Eye disorders) | 1 | 1 | 2 | 4
MYOPIA (Eye disorders) | 0 | 2 | 0 | 2
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 3 | 8 | 6 | 17
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 3 | 0 | 3
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 4 | 8 | 14
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 8 | 7 | 8 | 23
CONSTIPATION (Gastrointestinal disorders) | 3 | 5 | 5 | 13
DENTAL CARIES (Gastrointestinal disorders) | 2 | 1 | 0 | 3
DIARRHOEA (Gastrointestinal disorders) | 13 | 15 | 16 | 44
DYSPEPSIA (Gastrointestinal disorders) | 0 | 3 | 2 | 5
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 3 | 8 | 5 | 16
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 2 | 0 | 2 | 4
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 4 | 2 | 7
NAUSEA (Gastrointestinal disorders) | 7 | 5 | 6 | 18
TOOTH IMPACTED (Gastrointestinal disorders) | 0 | 3 | 0 | 3
TOOTHACHE (Gastrointestinal disorders) | 2 | 1 | 0 | 3
VOMITING (Gastrointestinal disorders) | 13 | 9 | 13 | 35
CHEST PAIN (General disorders) | 0 | 2 | 0 | 2
FATIGUE (General disorders) | 3 | 3 | 1 | 7
INFUSION SITE EXTRAVASATION (General disorders) | 2 | 1 | 0 | 3
PAIN (General disorders) | 4 | 2 | 0 | 6
PYREXIA (General disorders) | 9 | 5 | 5 | 19
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 | 1 | 2 | 3
HYPERSENSITIVITY (Immune system disorders) | 1 | 2 | 0 | 3
SEASONAL ALLERGY (Immune system disorders) | 0 | 1 | 3 | 4
BRONCHITIS (Infections and infestations) | 1 | 2 | 1 | 4
CELLULITIS (Infections and infestations) | 0 | 0 | 2 | 2
CROUP INFECTIOUS (Infections and infestations) | 1 | 0 | 2 | 3
EAR INFECTION (Infections and infestations) | 4 | 2 | 2 | 8
GASTROENTERITIS (Infections and infestations) | 4 | 5 | 2 | 11
GASTROENTERITIS VIRAL (Infections and infestations) | 4 | 3 | 2 | 9
GASTROINTESTINAL VIRAL INFECTION (Infections and infestations) | 2 | 0 | 2 | 4
INFECTIOUS MONONUCLEOSIS (Infections and infestations) | 0 | 2 | 1 | 3
INFLUENZA (Infections and infestations) | 3 | 7 | 4 | 14
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 0 | 0 | 2
OTITIS EXTERNA (Infections and infestations) | 2 | 0 | 1 | 3
OTITIS MEDIA (Infections and infestations) | 2 | 3 | 4 | 9
PARAINFLUENZAE VIRUS INFECTION (Infections and infestations) | 0 | 0 | 2 | 2
PHARYNGITIS (Infections and infestations) | 0 | 1 | 2 | 3
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 | 1 | 7 | 8
PNEUMONIA (Infections and infestations) | 1 | 1 | 2 | 4
POST PROCEDURAL INFECTION (Infections and infestations) | 0 | 3 | 0 | 3
RHINITIS (Infections and infestations) | 3 | 0 | 1 | 4
SINUSITIS (Infections and infestations) | 3 | 5 | 4 | 12
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 13 | 23 | 11 | 47
URINARY TRACT INFECTION (Infections and infestations) | 1 | 7 | 1 | 9
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 | 19 | 8 | 33
CONTUSION (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 3
FALL (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 4
HAND FRACTURE (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 3
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 4
STOMA SITE HYPERGRANULATION (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 2
BLOOD CHOLESTEROL INCREASED (Investigations) | 0 | 2 | 0 | 2
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 6 | 3 | 3 | 12
CARNITINE DECREASED (Investigations) | 3 | 0 | 1 | 4
ELECTROENCEPHALOGRAM ABNORMAL (Investigations) | 0 | 2 | 0 | 2
INFLUENZA A VIRUS TEST POSITIVE (Investigations) | 0 | 2 | 0 | 2
WEIGHT INCREASED (Investigations) | 0 | 3 | 1 | 4
ABNORMAL WEIGHT GAIN (Metabolism and nutrition disorders) | 0 | 3 | 0 | 3
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 1 | 2 | 4
DEHYDRATION (Metabolism and nutrition disorders) | 2 | 4 | 1 | 7
FLUID OVERLOAD (Metabolism and nutrition disorders) | 1 | 2 | 0 | 3
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 2 | 0 | 3
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 3 | 0 | 4
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2
HYPOPHAGIA (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2
OBESITY (Metabolism and nutrition disorders) | 0 | 3 | 1 | 4
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 4
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3 | 7
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 3
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 7
MYALGIA (Musculoskeletal and connective tissue disorders) | 7 | 8 | 2 | 17
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 | 3 | 7 | 14
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 10 | 18 | 6 | 34
HEADACHE (Nervous system disorders) | 5 | 3 | 5 | 13
HYPOTONIA (Nervous system disorders) | 2 | 1 | 0 | 3
LETHARGY (Nervous system disorders) | 1 | 0 | 2 | 3
MIGRAINE (Nervous system disorders) | 1 | 3 | 0 | 4
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 3 | 0 | 4
ANXIETY (Psychiatric disorders) | 6 | 4 | 1 | 11
ATTENTION DEFICIT/HYPERACTIVITY DISORDER (Psychiatric disorders) | 1 | 2 | 1 | 4
DEPRESSION (Psychiatric disorders) | 1 | 3 | 0 | 4
ENURESIS (Psychiatric disorders) | 2 | 0 | 0 | 2
INSOMNIA (Psychiatric disorders) | 1 | 3 | 0 | 4
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 | 5 | 0 | 5
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 6 | 15
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 5
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 3 | 9
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 3 | 8
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 9 | 3 | 13
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 5
ACNE (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 5
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 3
DERMATITIS DIAPER (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 3
RASH (Skin and subcutaneous tissue disorders) | 5 | 3 | 3 | 11
HYPERTENSION (Vascular disorders) | 1 | 6 | 0 | 7
POOR VENOUS ACCESS (Vascular disorders) | 3 | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT02214160/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/60/NCT02214160/SAP_001.pdf